CLINICAL TRIAL: NCT06395441
Title: Phase III Study of Ginseng for Cancer Related Fatigue
Brief Title: Wisconsin Ginseng for Decreasing Cancer Related Fatigue
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MC231004; NCI-2024-03375 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23-012122 (Other: Mayo Clinic Institutional Review Board); MC231004 (Other: Mayo Clinic in Rochester); MNCCTN037 (Other: MN Cancer Clinical Trials Network)
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Malignant Solid Neoplasm
MeSH Terms: interventions — Asian ginseng

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Research staff, other than pharmacy, are blinded, and will dispense product to the patient. Option to unblind: At the end of treatment, if, in the judgment of patient or patient's attending clinician, it would be helpful for the future of patient's clinical care, the code may be broken.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (Western ginseng) (Experimental): Patients receive Western ginseng PO BID on days 1-56. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Dietary Supplement: American Ginseng; Other: Questionnaire Administration
- Group II (placebo) (Placebo Comparator): Patients receive placebo PO BID on days 1-56. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Placebo Administration; Other: Questionnaire Administration

INTERVENTIONS:
Dietary Supplement: American Ginseng — Given PO
  Other Names: Ginseng; Ginseng Root; Panax quinquifolius
  Arms: Group I (Western ginseng)
Drug: Placebo Administration — Given PO
  Arms: Group II (placebo)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase III trial compares the effect of Wisconsin ginseng (panax quinquefolius) to placebo in patients with cancer that suffer from significant fatigue. Fatigue is among the most challenging symptoms to manage in patients with cancer, both on or off active treatment. This symptom complex meaningfully contributes to psychosocial distress, healthcare costs, and it also interferes with the delivery of anticancer therapies. American ginseng (Western ginseng) appears to be a promising appearing agent for treating cancer related fatigue. Western ginseng may reduce cancer-related fatigue.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the efficacy of ginseng as assessed by a single item measure of fatigue at 8 weeks.

SECONDARY OBJECTIVES:

I. To estimate changes in fatigue via the single item measure of fatigue from baseline to week 4, the Global Impression of Change at week 4 and 8, and the Functional Assessment of Chronic Illness Therapy-Fatigue Scale (FACIT-Fatigue) at week 4 and 8.

II. To evaluate the frequency and severity of toxicity as reported by the patient on the Ginseng Symptom Experience Diary where patients rate (on a 0 to 10 scale) their toxicities experienced while on study.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients receive Western ginseng orally (PO) twice daily (BID) on days 1-56.

GROUP II: Patients receive placebo PO BID on days 1-56.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Has received or is receiving treatment for a solid-organ malignancy (not hematologic)
* History of cancer-related fatigue as defined by an average score ≥ 4 over the past 30 days on the numeric analogue scale. Patients can answer questions orally rather than completing worksheet
* Baseline control of insomnia: Insomnia ≤ 4 on Linear Analogue Scale. Patients can answer questions orally rather than completing worksheet
* Baseline control of pain: Pain ≤ 4 on Linear Analogue Scale. Patients can answer questions orally rather than completing worksheet
* Life expectancy ≥ 6 months
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Hemoglobin ≥ 10.0 g/dL (patients must not have been transfused in the preceding 90 days to meet this criterion) (≤ 180 days prior to registration)
* Alanine aminotransferase (ALT) or aspartate transaminase (AST) ≤ 3 x upper limit normal (ULN) (≤ 180 days prior to registration)
* Creatinine ≤ 1.5 x ULN (≤ 180 days prior to registration)
* No clinical suspicion of hypothyroidism within 180 days prior to registration [if clinical suspicion of hypothyroidism exists, a documented thyroid stimulating hormone (TSH) < 5 milli-international units per liter (mIU/L) is required]
* Negative pregnancy test done ≤ 7 days prior to registration, for persons of childbearing potential only
* Ability to complete questionnaire(s) by themselves or with assistance
* Provide informed consent

Exclusion Criteria:

* Any known hypersensitivity to ginseng
* Currently using any other pharmacologic agents to specifically treat fatigue including psychostimulants or antidepressants. Note: Antidepressants used to treat items other than fatigue (such as hot flashes or depression) are allowed if the patient has been on a stable dose for ≥ 30 days and plan to continue such for 8 weeks. Exercise is allowed
* Psychiatric disorder such as poorly controlled depression, manic depressive disorder, obsessive compulsive disorder, or schizophrenia (defined per medical history)
* Use of erythropoietic agents ≤ 6 months
* Uncontrolled hypertension on more than three occasions (diastolic blood pressure ≥ 100, systolic ≥ 160) measured ≤ 180 days prior to randomization
* Surgery that required general anesthetic ≤ 30 days prior to randomization
* Malnutrition, active infection, severe depression, or significant pulmonary disease and cardiovascular disease (as determined by the attending clinician), as they could impact fatigue
* Use of any over the counter herbal/dietary supplement marketed for fatigue or energy (for example, products containing any type of ginseng, Rhodiola rosea, guarana, or anything called an "adaptogen")
* Currently using an antidiabetic drug, warfarin or monamine oxide inhibitor
* Treating provider anticipates a change to the anti-cancer treatment program in the next 8 weeks (i.e., the intervention period)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change in fatigue | Baseline to 8 weeks
  Will be measured by the Linear Analog Scale for Fatigue, a single-item questionnaire rating fatigue over the pats week on a scale of 0-10 where 0=no fatigue at all and 10=fatigue as bad as it can be.

SECONDARY OUTCOMES:
Change in fatigue | Baseline, 4 and 8 weeks
  Will be measured by the Functional Assessment of Chronic Illness Therapy- Fatigue (FACIT-Fatigue) Scale, which consists of 13 questions answered on a scale of 0-4 where 0=not at all and 4=very much.
Percentage of patients who perceive moderate to very much better fatigue | At 8 weeks
  Will be measured by the Global Impression of Change, which consists of 3 questions answered on a scale of -3 (very much worse) to 3 (very much better), one question as to whether the participants thought they were receiving the intervention (ginseng) or placebo, and one question related to satisfaction with the effect of the treatment on their fatigue (yes/no).
Incidence of adverse events | Up to 8 weeks
  Will be measured by the Common Terminology Criteria for Adverse Events (CTCAE) and/or the Ginseng Symptom Experience Diary and compared between arms.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S. Childs, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (15):
- United States (15):
  - Mayo Clinic Health System in Albert Lea, Albert Lea, Minnesota
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Essentia Health Deer River Clinic, Deer River, Minnesota
  - Essentia Health St. Mary's Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Fosston, Fosston, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Mayo Clinic Health System-Mankato, Mankato, Minnesota
  - MMCORC CentraCare Monticello Cancer Center, Monticello, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Sanford Worthington Medical Center, Worthington, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials